CLINICAL TRIAL: NCT03331562
Title: A SU2C Catalyst ® Randomized Phase II Trial of the PD1 Inhibitor Pembrolizumab With or Without a Vitamin D Receptor Agonist Paricalcitol in Patients With Stage IV Pancreatic Cancer Who Have Been Placed in Best Possible Response
Brief Title: A SU2C Catalyst® Trial of a PD1 Inhibitor With or Without a Vitamin D Analog for the Maintenance of Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Genomics Research Institute (Other)
Collaborators: Stand Up To Cancer (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGen 17-001; MISP# 56240 (Other: Merck Sharp & Dohme Corp. a Subsidiary of Merck & Co., Inc.)
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer; Pancreas Adenocarcinoma; Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma
Keywords: Pembrolizumab; Paricalcitol; Pancreatic cancer; Metastatic Pancreatic Cancer; Vitamin D Receptor (VDR); Immune Checkpoint Inhibitor; VDR agonist; PD1 Inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; paricalcitol

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled phase II trial with the identity of the treatment unknown to the patients, investigators, and the Sponsor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- pembrolizumab & paricalcitol (Active Comparator): pembrolizumab 200 mg IV q 3 weeks and paricalcitol 25 mcg IV 3 xs per week
  Interventions: Drug: Pembrolizumab; Drug: paricalcitol
- pembrolizumab & placebo (Placebo Comparator): pembrolizumab 200 mg IV q 3 weeks & placebo- normal saline IV 3 xs per week
  Interventions: Drug: Pembrolizumab; Drug: placebo

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab solution for infusion
  Other Names: Keytruda
Drug: paricalcitol — Paricalcitol solution for injection
  Other Names: Zemplar
  Arms: pembrolizumab & paricalcitol
Drug: placebo — normal saline solution for injection
  Other Names: placebo for paricalcitol
  Arms: pembrolizumab & placebo

SUMMARY:
Chemotherapy regimens for pancreatic cancer can now stabilize a patient's cancer and/or place some patients in remission or partial remission. The challenge now is to find options for maintenance therapies that will improve survival and allow continued benefits with minimal toxicities and inconvenience to the patients. This study will determine the effects of one possible maintenance regimen.

The study is being conducted to determine the effects that pembrolizumab with or without the addition of paricalcitol may have on pancreatic cancer. Half of the patients will be randomized to receive pembrolizumab + paricalcitol and half to receive pembrolizumab + placebo.

DETAILED DESCRIPTION:
Pembrolizumab (also known as Keytruda®), which is approved in the USA and some other countries, is available by prescription to treat several different cancers, but has not been approved to treat pancreatic cancer. Pembrolizumab helps the body detect and fight cancer by making cancer cells more vulnerable to attack by the body's immune system. This medication binds to and lessens the action of specific parts of cells in the body's immune system, which act to modulate or balance the immune response. By decreasing this modulation of the immune response, the body's own system may be better able to fight the cancer. Pembrolizumab is known as an immune checkpoint inhibitor.

It is thought that the effect of pembrolizumab could possibly be strengthened by the addition of paricalcitol, which is a form of vitamin D. Paricalcitol may make the cells in the immune system more sensitive to the activity of pembrolizumab and could make the local environment hostile to the cancer cells. Both activities could be effective against cancer growth.

Paricalcitol (also known as Zemplar®) is used to treat high levels of parathyroid hormone and prevent bone loss in patients with advanced kidney disease. Paricalcitol is not approved by the FDA for the treatment of advanced pancreatic cancer.

The effects of the study drugs will be assessed by repeated radiological imaging (CT scans), incidence of adverse reactions, and survival rates.

Participants will also be asked to provide biological specimens for the study team to measure cellular changes. This will include fecal matter (stool), blood, and tumor tissue.

The Food and Drug Administration (FDA) has determined that this study meets the requirements for Investigational New Drug (IND) Exemption.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Histologically or cytologically confirmed pancreatic adenocarcinoma with metastasis, who had obtained a best response of at least stable disease (SD) or a partial response (PR) for a period of 2 months with no further shrinkage of ≥ 30% on scan on their first line of chemotherapy for their advanced metastatic disease. Note: Patients that have had prior chemotherapy as adjuvant or neoadjuvant therapy are permitted.
4. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
5. Able to submit an archival tumor specimen (primary or metastatic site) and a discussion is documented with trial investigator at screening that patient will consider providing tissue from a newly obtained core or excisional biopsy of a tumor lesion at baseline and a second biopsy 9 weeks after starting trial treatment, unless tumor is considered inaccessible or biopsy is otherwise considered not in the patients best interest. Participation in this trial is not contingent on patient consenting to optional tumor biopsies.
6. Demonstrate adequate organ function as defined in protocol, AND serum corrected calcium value must be ≤ Institutional Upper Limit of Normal (ULN) and ≥ 8.0 mg/dL, and phosphorus levels must be ≤ Institutional ULN and ≥ 2.5 mg/dL.
7. Female participants of childbearing potential should have a negative serum pregnancy test within 24 hours prior to receiving first dose of trial medication.
8. A female participant is eligible to participate if she is not pregnant , not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in protocol

      OR
   2. A WOCBP who agrees to follow the contraceptive guidance in protocol during the treatment period and for at least 120 days after the last dose of trial treatment.
9. Male participants must agree to use a contraception as detailed in protocol during the treatment period and for at least 120 days after the last dose of trial treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Is currently participating and receiving trial therapy or has participated in a trial of an investigational agent and received trial therapy or used an investigational device within 4 weeks of the first dose of trial treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
3. Has a known history of active TB (Mycobacterium tuberculosis).
4. Hypersensitivity to pembrolizumab or paricalcitol or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1/Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle1/ Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent(s).

   Note: Patients with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the trial.

   Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Has a serum vitamin D level of ≥ 50 ng/mL
16. Currently taking a strong cytochrome P450 3A (CYP3A) inhibitors that cannot be discontinued prior to trial enrollment and for the duration of trial. This includes but is not is limited to: boceprevir clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has a known history of or is positive for Hepatitis B (e.g., HBsAg reactive) or Hepatitis C virus (e.g., HCV RNA [qualitative] is detected).

    Note: Without known history testing needs to be performed to determine eligibility.
19. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator, or patient receiving a digitalis derivative.
20. Has received a live vaccine within 30 days of planned start of trial therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Von Hoff, MD, FACS, Study Director — Translational Genomics Research Institute (TGen) An Affiliate of City of Hope
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Atlantic Medical Group-Oncology Morristown Medical Center, Morristown, New Jersey
  - Baylor University Medical Center Charles A. Sammons Cancer Center, Dallas, Texas
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung V, Alistar A, Becerra C, Kasi A, Borazanci E, Jameson GS, Roe DJ, Wertheim BC, Cridebring D, Truitt M, Downes M, Barrett MT, Korn R, Lee K, Han H, Evans R, Von Hoff DD. Pembrolizumab +/- paricalcitol in metastatic pancreatic cancer postmaximal cytoreduction. Oncologist. 2025 Jan 17;30(1):oyae323. doi: 10.1093/oncolo/oyae323. PMID 39846984

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Started (Randomized to study arm, received allocated study treatment) | 12 | 12
Completed (Patients continued on study treatment until disease progression) | 9 | 12
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Full Range); unit: years] | 63.8 [42.9 to 77.9] | 69.3 [50.5 to 76.7] | 67.6 [42.9 to 77.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG performance) status scales and criteria are used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  ECOG 0=Fully active, able to carry on all pre-disease performance without restriction
  ECOG=1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG 0 | 5 | 4 | 9
    ECOG 1 | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression- Free Survival at 6 Months From Initiation of Trial Treatment
Description: Progression Free Survival (PFS) defined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) survival in the absence of death or progressive disease which is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 6 months from trial treatment initiation cycle 1/day 1. Each treatment cycle is 21 days.
Population: All patients that receive trial treatment will be included in the analysis. Excludes 3 participants in the pembrolizumab + paricalcitol group: 1 participant that died due to other cause before 6 months, 2 participants who withdrew from study treatment before 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 9 | 12
Participants | 0 | 2
Statistical Analysis 1: Comparison: Pembrolizumab & Placebo; Test type: Superiority; p = .31, Fisher Exact; Risk Ratio (RR) = 0, 95% CI 1-sided [lower limit 0] — Lower bound cannot be estimated because there were 0 events in the comparison group

2. Secondary Outcome: Incidence of Treatment-related Toxicities as Assessed by CTCAE v4.0 From cycle1/Day 1 Through 30 Days After the Last Dose of Trial Treatment.
Description: All adverse events occurring on or after Cycle 1/day 1through 30 days after the last dose of trial treatment will be summarized by body systems and per grade according to NCI-CTCAE Version 4.
Time Frame: initiation of trial treatment cycle 1/day 1 through 30 days after last dose of trial treatment. Each treatment cycle is 21 days.
Population: All patients who received any amount of trial treatment were included in the analysis. The reported AEs are those noted as possibly or definitely related to study agents.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Abdominal bloating | 1 | 0
  Abdominal pain | 1 | 2
  ALT increase | 2 | 0
  Alkaline phosphatase increase | 1 | 0
  Anemia | 0 | 1
  Arthralgia | 2 | 0
  AST increase | 2 | 1
  Creatinine increase | 2 | 0
  Hypertension | 0 | 2
  Hypophysitis | 1 | 0
  Nausea | 1 | 0
  Pruritis | 1 | 0
  Uticaria | 0 | 1
  Vomiting | 1 | 0

3. Secondary Outcome: Difference in Overall Survival (OS) in Patients Administered the Combination of Paricalcitol Plus Pembrolizumab Versus Pembrolizumab Alone
Description: Duration of survival will be defined as the time from initial treatment (cycle1/day1) until death. Overall survival will be estimated for each arm using a Kaplan-Meier estimate.
Time Frame: From date of treatment initiation cycle 1/day 1 until death from any cause, assessed up to 24 months ( the end of the study).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 12 | 12
months | 10.4 [2.9 to NA] — The upper bound of the confidence interval cannot be calculated because the upper bound did not fall below 50% by the end of the study. | NA [2.5 to NA] — Median OS not be calculated for the pembrolizumab & placebo group because the median has not yet been reached (only 4 deaths of 12 participants). The upper bound of the confidence interval cannot be calculated because the upper bound did not fall below 50% by the end of the study.

4. Secondary Outcome: Change in Tumor Mutational Landscape and Transcriptional Programs Using Unbiased Genome-wide Sequencing
Description: Mutational landscapes, transcriptional programs in tumor tissue
Time Frame: Optional tumor biopsy taken at baseline and at 9 +/- 1 week following initiation of treatment
Population: Data could not be analyzed due to lack of funding for the project.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cellular VDR Targets in the Immune Microenvironment With PD1 Blockade
Description: Identify cellular VDR targets in the immune microenvironment
Time Frame: From baseline, at 9 +/- 1 week following initiation of treatment, at the time of confirmed response, and at the time of trial treatment discontinuation for any reason, up to 24 months ( 35 treatment cycles).
Population: Due to lack of funding, this analysis could not be performed.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Exploratory: Difference in Disease Progression According to RECIST 1.1 and iRECIST
Description: Difference in disease progression according to RECIST 1.1 and iRECIST criteria
Time Frame: tumor assessments performed every 9 +/- 1 week while on treatment, up to 24 months.
Population: This planned analysis was not performed, as we were not able to obtain confirmation of disease progression by iRECIST for a majority of the patients.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Exploratory: Utility of a Patient Personalized Clinical Benefit (PPCB) Phone Based Application
Description: Patient compliance rate of completing the PPCB application was calculated by the total percentage of completed questionnaires over expected questionnaires across all participants.
Time Frame: From baseline, patients will complete the PPCB App weekly during trial treatment, and at the time of trial treatment discontinuation for any reason, assessed up to 24 months (35 treatment cycles).Each treatment cycle is 21 days.
Population: All patients were included in the analysis.
Measure: Number; unit: % of questionnaires completed
Groups:
- Pembrolizumab & Paricalcitol: Compliance rate for all participants treated in the Pembrolizumab & Paricalcitol arm
- Pembrolizumab & Placebo: Compliance rate for all participants treated in the Pembrolizumab & Placebo Arm
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 12 | 12
% of questionnaires completed | 89.4 | 92.8

8. Other Pre Specified Outcome: Exploratory:Improvement in Symptoms as Recorded by the Patient Personalized Clinical Benefit (PPCB) With Progression at 6 Months by RECIST 1.1
Description: Improvement in symptoms as recorded by the Patient Personalized Clinical Benefit (PPCB)
Time Frame: From baseline, patients will complete the PPCB App weekly during trial treatment, and at the time of trial treatment discontinuation for any reason, assessed up to 24 months (35 treatment cycles). Each treatment cycle is 21 days.
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab & Paricalcitol: All participants that completed the questionnaires in Pembrolizumab & Paricalcitol arm
- Pembrolizumab & Placebo: All participants who completed questionnaire in Pembrolizumab & Placebo Arm
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Improvement in symptoms | 8 | 7
  Worsening in symptoms | 4 | 3
  No change in symptoms | 0 | 2

9. Other Pre Specified Outcome: Changes in Tumor and/or Tissue Texture on Imaging in Both Arms of the Trial Using Quantitative Textural Analysis (QTA)
Description: Differences in tumor and/or tissue texture on CT scans between the two treatment arms
Time Frame: tumor assessments performed every 9 +/- 1 week while on treatment, up to 24 months.
Population: Due to lack of funding analysis could be be completed.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Exploratory: Monitor and Compare the Gut Microbial Communities in Both Arms of the Trial
Description: Differences in gut microbial communities within and between fecal samples using alpha and beta diversity metrics based on 16S rRNA sequencing
Time Frame: Fecal swab samples collected pre and post dose day 1 of each cycle, up to 35 treatment cycles. Each treatment cycle is 21 days.
Population: Due to lack of funding analysis could be be completed.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of treatment allocation/randomization through 30 days following cessation of study treatment.
Description: Participants with multiple events for a given AE term were counted only once for each AE term. If the same AE term was reported more than once for a participant, only the AE term with the highest grade was included.
Arm/Group | Pembrolizumab & Paricalcitol | Pembrolizumab & Placebo
All-Cause Mortality (participants affected / at risk) | 8/12 | 4/12
Serious Adverse Events (participants affected / at risk) | 4/12 | 4/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab & Paricalcitol (N=12) | Pembrolizumab & Placebo (N=12)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, hepatorenal syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, takotsubo cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Malignant Neoplasms- Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab & Paricalcitol (N=12) | Pembrolizumab & Placebo (N=12)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - other, cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorders - other, hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Bloating (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorder other: bleeding with stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Other- cold sensitivity (General disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders other: biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Other, neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Other- ammonia increased (Investigations) | 1 (1) | 0 (0)
Other, lactic acid increased (Investigations) | 1 (1) | 0 (0)
Other, thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Other, temporomandibular joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flash (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to lack of grant funding, the other exploratory objectives to assess the changes in tumor and/or tissue texture on imaging, and to monitor and compare gut microbial communities in both arms, have not yet been able to be accomplished. The Investigators are looking for some way to fund the exploratory objectives in the future.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT03331562/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03331562/SAP_001.pdf